CLINICAL TRIAL: NCT02187211
Title: Minocycline's Effects on Alcohol Responses in Humans
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 1312013129; 1R21AA023150-01A1 (NIH)
Record Dates: First submitted 2014-07-08; First posted 2014-07-10 (Estimated); Last update posted 2020-03-09 (Actual); Status verified 2020-03

CONDITIONS: Alcohol Dependence
Keywords: Alcohol Dependence; Minocycline
MeSH Terms: conditions — Alcoholism; cyclopia sequence | interventions — Minocycline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Minocycline Low Dose (Experimental): Participants in this arm will receive a low dose (200mg/day) of Minocycline for 10 days
  Interventions: Drug: Minocycline
- Minocycline High Dose (Experimental): Participants in this arm will receive a high dose (400mg/day) of Minocycline for 10 days
  Interventions: Drug: Minocycline
- Placebo (Placebo Comparator): Participants in this arm will receive the Placebo for 10 days
  Interventions: Drug: Placebo (for Minocycline)

INTERVENTIONS:
Drug: Minocycline
  Arms: Minocycline High Dose; Minocycline Low Dose
Drug: Placebo (for Minocycline)
  Arms: Placebo

SUMMARY:
This is a double-blind, placebo-controlled, outpatient study with a between-groups design. Sixty male and female heavy social drinkers will be randomly assigned to minocycline (200 or 400 mg/day) or placebo for 10 days. In the first 7 days of treatment, subjects will have 3 outpatient visits for medication administration, dispensing of take-home doses and monitoring of any adverse effects from study medications. On days 8 and 10 of treatment, subjects will have 2 laboratory sessions where alcohol or placebo will be administered intravenously using a clamp procedure. Alcohol administration will use a breath alcohol concentration (BrAc) method, targeting 100 mg %. The alcohol clamp procedure will allow collection of multiple outcome measures including subjective, motor, cognitive measurement and plasma cytokine levels.

ELIGIBILITY:
Inclusion Criteria:

1. Male and females, between the ages of 21 and 50;
2. Heavy social drinkers who are defined as consuming ≥10 standard alcoholic drinks per week with one to five weekly "binge" drinking episodes, (5 plus drinks per occasion for men; 4 plus drinks for women). No maximum level of alcohol consumption will be defined a priori but individuals who met current DSM -IV criteria for AUD will be excluded from the study;
3. No current drug use disorder of any drugs of abuse (except alcohol and tobacco);
4. No current medical problems and normal ECG; 5) For women, not pregnant as determined by pregnancy screening nor breast feeding, and using acceptable birth control methods.

Exclusion Criteria:

1. Current major psychiatric illnesses including mood, psychotic, or anxiety disorders;
2. History of major medical illnesses; including liver diseases, heart disease, chronic pain or other medical conditions that the physician investigator deems contraindicated for the subject to be in the study;
3. Liver function tests (ALT or AST) greater than 3 times normal;
4. Allergy to minocycline or other tetracyclines;
5. Participants who at any appointment have a Clinical Institute Withdrawal Assessment Scale (CIWA) [36, 37] score of 4 or greater, or who report any history of alcohol withdrawal within the past 6 months.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
Biphasic Alcohol Effects Scale (BAES) | Days 1-10
  BAES will be used to measure the stimulant and sedative effects of alcohol during the test sessions. This instrument has been found to be a sensitive and reliable measure to study medication influences on alcohol effects

CONTACTS AND LOCATIONS:
Overall Officials: Ismene Petrakis, M.D., Principal Investigator — Yale University
Locations (1):
- VA Connecticut Healthcare System, West Haven, Connecticut, United States